CLINICAL TRIAL: NCT02348203
Title: Clinical Study of the Effect of Combined Treatment of Aspirin and Zileuton on Biomarkers of Tobacco-Related Carcinogenesis in Current Smokers
Brief Title: Aspirin and Zileuton and Biomarker Expression in Nasal Tissue of Current Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCI-2015-00061; NCI-2015-00061 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00031; 1403269898 (Other: Banner University Medical Center - Tucson); UAZ2013-02-01 (Other: DCP); N01CN00031 (NIH); P30CA023074 (NIH)
Record Dates: First submitted 2015-01-27; First posted 2015-01-28 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Aspirin; zileuton

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (aspirin, zileuton) (Experimental): Patients receive aspirin PO QD and zileuton PO BID for 12 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: Aspirin; Other: Laboratory Biomarker Analysis; Drug: Zileuton
- Arm II (double placebo) (Placebo Comparator): Patients receive aspirin placebo PO QD and zileuton placebo PO BID for 12 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration

INTERVENTIONS:
Drug: Aspirin — Given PO
  Other Names: Acetylsalicylic Acid; ASA; Aspergum; Ecotrin; Empirin; Entericin; Extren; Measurin
  Arms: Arm I (aspirin, zileuton)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given aspirin placebo PO
  Arms: Arm II (double placebo)
Other: Placebo Administration — Given zileuton placebo PO
  Arms: Arm II (double placebo)
Drug: Zileuton — Given PO
  Other Names: Zyflo
  Arms: Arm I (aspirin, zileuton)

SUMMARY:
This randomized phase II trial studies the effects of aspirin and zileuton on genes related to tobacco use in current smokers. Aspirin and zileuton may interfere with genes related to tobacco use and may be useful in preventing lung cancer in current smokers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To analyze the impact of combined treatment of acetylsalicylic acid (ASA) (aspirin) and zileuton on smoking-related gene expression signature in the nasal epithelium in current smokers and to analyze any difference between the ASA and zileuton intervention and placebo control.

SECONDARY OBJECTIVES:

I. To assess the impact of ASA and zileuton on three lung cancer gene signatures (an 80-gene bronchial signature, a phosphatidylinositol 3-kinase [PI3K] pathway gene signature and a nasal diagnostic gene signature) and to compare this to placebo control.

II. To determine whether the change in the smoking-related gene expression signature and the three lung cancer gene signatures of nasal epithelium persists 10-14 days off agent intervention.

III. To measure urinary prostaglandin E metabolite (PGE-M) and leukotriene E(4) (LTE[4]) levels in current smokers after ASA and zileuton.

IV. To assess the safety in current smokers of 12 week exposure to ASA and zileuton.

V. To evaluate a gender effect in the modulatory effects of ASA and zileuton on smoking related-gene expression signature.

VI. To explore the effect of ASA and zileuton on the metabolomics profile of the arachidonic acid pathway.

VII. To explore, in a discovery-driven fashion, the effect of ASA and zileuton on whole-genome gene expression.

VIII. To analyze the impact of ASA and zileuton on karyometric analysis of buccal cells.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive aspirin orally (PO) once daily (QD) and zileuton PO twice daily (BID) for 12 weeks in the absence of unacceptable toxicity.

ARM II: Patients receive aspirin placebo PO QD and zileuton placebo PO BID for 12 weeks.

After completion of study treatment, patients are followed up for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Current tobacco smokers with >= 20 pack years of self-reported smoking exposure and an average use of >= 10 cigarettes/day
* Karnofsky >= 70%
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Hematocrit >= the lower institutional limit
* Platelets >= the lower institutional limits
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) within normal institutional limits
* Creatinine =< the upper institutional limits
* Prothrombin time (PT)/partial thromboplastin time (PTT) within normal institutional limits
* Fertile subjects must use adequate contraception (abstinence, barrier methods, or birth control pills) prior to study entry and for the duration of study participation; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Participants may have a history of indeterminate pulmonary nodule(s) by chest imaging if nodule follow-up has been completed or the study procedures would not interfere with nodule follow-up
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of allergic reaction to aspirin or attributed to compounds of similar chemical or biologic composition to aspirin, including other nonsteroidal anti-inflammatory drugs (NSAIDs)
* Gastric intolerance attributable to ASA or NSAIDs
* History of gastric ulcer within the past 5 years (with or without bleeding)
* Use of ASA or NSAIDs for more than 5 days per month within 3 months of enrollment
* Not willing or are unable to refrain from use of any non-study ASA, NSAIDs and leukotriene antagonists during the study period
* Adult asthma
* Chronic, current or recent (within the past three months) use of leukotriene antagonists
* Require chronic anticoagulation or anti-platelet therapy
* History of bleeding disorder or hemorrhagic stroke
* Chronic, current or recent (within the past three months) use of glucocorticoids (systemic, topical and/or nasal sprays or steroid topical creams to large body surface area); use of steroid topical creams for small body areas (=< 10% body surface) during study intervention is allowed
* History of chronic sinusitis or recent nasal polyps
* History of, or current, active or chronic liver disease even if transaminases have normalized
* History of allergic reaction to zileuton or attributed to compounds of similar chemical or biologic composition to zileuton
* Are taking drugs known to interact with zileuton, including theophylline, warfarin, and propranolol
* Not willing or are unable to limit alcohol consumption to =< 2 alcoholic beverages a day during the study period
* Pregnant or lactating women; breastfeeding should be discontinued if the mother is treated with aspirin; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Participants may not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Have a known history of inability to absorb an oral agent
* Invasive cancer within the past five years except non-melanoma skin cancer
* Urine cotinine level, if collected at screening, does not confirm active smoking status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda L Garland, Principal Investigator — The University of Arizona Medical Center-University Campus
Locations (2):
- United States (2):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Boston University School of Medicine, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Started | 31 | 32
Completed | 21 | 22
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo) | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (8.6) | 53.5 (10.7) | 51.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 28 | 24 | 52
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Changes in a Smoking-related Gene Expression Signature Score in the Nasal Epithelium of Current Smokers
Description: Change in a nasal smoking-related gene expression signature score derived from prior research was compared between the two study arms. Prior research showed that a higher score was observed in never smokers compared to current smokers. An increased score implicated a more favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 12 weeks (End-of-intervention)
Population: The number of participants analyzed is different from the numbers provided in the Participant Flow Module because gene expression analysis was restricted to samples that met quality metrics.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 19 | 21
score on a scale | -0.15 (2.89) | 0.26 (2.26)

2. Secondary Outcome: Changes in Three Lung Cancer Gene Signatures (an 80-gene Bronchial Signature, a PI3K Pathway Gene Signature and a Nasal Diagnostic Gene Signature) in the Nasal Epithelium of Current Smokers
Description: Change in three lung cancer gene signatures (an 80-gene bronchial signature, a PI3K pathway gene signature and a nasal diagnostic gene signature) derived from prior research was compared between the two study arms. A decreased signature score implicated a more favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 12 weeks (End of Intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 19 | 21
score on a scale
  bronchial smoking signature | -1.0 (2.87) | -0.43 (3.37)
  PI3 pathway gene signature | -0.32 (1.57) | 0.42 (1.68)
  nasal diagnostic gene signature | 1.82 (8.63) | 2.17 (11.21)

3. Secondary Outcome: Changes in a Smoking-related Gene Expression Signature Score in the Nasal Epithelium of Current Smokers 10-14 Days Post Intervention
Description: Change (from baseline to 10-14 days off intervention) in a nasal smoking-related gene expression signature score derived from prior research was compared between the two study arms. Prior research showed that a higher score was observed in never smokers compared to current smokers. An increased score implicated a more favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 14 days post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 19 | 21
score on a scale | -0.24 (3.04) | -1.16 (3.55)

4. Secondary Outcome: Changes in Three Lung Cancer Gene Signatures (an 80-gene Bronchial Signature, a PI3K Pathway Gene Signature and a Nasal Diagnostic Gene Signature) in the Nasal Epithelium of Current Smokers 10-14 Days Post Intervention
Description: Change (from baseline to 10-14 days off intervention) in three lung cancer gene signatures (an 80-gene bronchial signature, a PI3K pathway gene signature and a nasal diagnostic gene signature) derived from prior research was compared between the two study arms. A decreased signature score implicated a more favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 14 days post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 19 | 21
score on a scale
  bronchial signature | -1.37 (2.69) | 0.88 (3.71)
  PI3K pathway gene signature | -0.16 (1.63) | 0.71 (2.35)
  nasal diagnostic gene signature | 2.78 (6.35) | -1.98 (11.58)

5. Secondary Outcome: Change in Urinary PGE-M Levels
Time Frame: Baseline to 12 weeks (End-of-intervention)
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 21 | 22
ng/mg creatinine | -5.9 (13.9) | 0.71 (9.3)

6. Secondary Outcome: Change in Urinary LTE (4) Levels
Time Frame: Baseline to 12 weeks (End-of-intervention)
Measure: Mean (Standard Deviation); unit: pg/mg creatinine
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 21 | 22
pg/mg creatinine | -57.6 (65.6) | 35.2 (92.7)

7. Secondary Outcome: Number of Participants Experiencing Possibly/Probably/Definitely-related Adverse Events
Time Frame: Up to 2 weeks post-treatment
Population: All participants who have received at least one dose of the study agent.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 31 | 32
Participants | 9 | 8

8. Secondary Outcome: Gender Effect on Smoking-related Gene Expression Signature
Description: Change in a nasal smoking-related gene expression signature score derived from prior research was analyzed by gender. Prior research showed that a higher score was observed in never smokers compared to current smokers. An increased score implicated a more favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 12 weeks (End-of-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 19 | 21
score on a scale
  Females: number analyzed (Participants) | 8 | 11
  Females | 0.01 (2.93) | -0.20 (2.01)
  Males: number analyzed (Participants) | 11 | 10
  Males | -0.27 (2.99) | 0.76 (2.51)

9. Secondary Outcome: Changes in the Metabolomics Profile of the Arachidonic Acid Pathway
Description: Two sample t tests will be performed to evaluate whether or not there are significant differences in changes in oxylipin metabolome between the treatment and placebo groups. In addition, system biology methods will also be used to analyze the oxylipin metabolome data.
Time Frame: Baseline to 12 weeks (End-of-intervention)
Population: Data were not collected.
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Genes Differentially Expressed After Aspirin and Zileuton Intervention Compared to Placebo
Description: Number of genes differentially expressed after aspirin and zileuton intervention compared to placebo using whole-genome gene expression data
Time Frame: Baseline to 12 weeks (End-of-intervention)
Measure: Number; unit: gene
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 19 | 21
gene | 83 | 0

11. Secondary Outcome: Impact of ASA and Zileuton on Karyometric Analysis of Buccal Cells
Time Frame: Up to week 12
Population: Data were not collected.
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time that the first dose of study drug was taken until 2 weeks after participants come off the 12-week agent intervention.
Arm/Group | Arm I (Aspirin, Zileuton) | Arm II (Double Placebo)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 25/31 | 17/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Aspirin, Zileuton) (N=31) | Arm II (Double Placebo) (N=32)
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Weight gain (Investigations) | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 4 | 2
Flu like symptoms (General disorders) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Weight loss (Investigations) | 0 | 2
Hypertension (Vascular disorders) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT02348203/Prot_SAP_000.pdf